CLINICAL TRIAL: NCT02724098
Title: Bioavailability of Subcutaneously Given Dexmedetomidine in Healthy Volunteers
Brief Title: Bioavailability of Subcutaneous Dexmedetomidine
Acronym: ScDex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T30/2016
Record Dates: First submitted 2016-02-12; First posted 2016-03-31 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Pain
Keywords: Palliative Therapy
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous (Active Comparator): 1 µg/kg dexmedetomidine (dexmedetomidine hydrochloride 100 microg/ml, Dexdor® Orion Oyj, Espoo, Finland) diluted in 10 ml of sodium chloride will be administered intravenously in 10 min at a constant rate using an infusion pump.
  Interventions: Drug: Dexmedetomidine
- subcutaneous (Active Comparator): 1 µg/kg dexmedetomidine (dexmedetomidine hydrochloride 100 microg/ml, Dexdor® Orion Oyj, Espoo, Finland) will be administered subcutaneously undiluted.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
The aim of this study is to investigate the pharmacokinetics of subcutaneously administered dexmedetomidine in healthy volunteers. The absolute bioavailability of subcutaneously administered dexmedetomidine will be calculated. In addition, the investigators will report the effects of subcutaneously administered dexmedetomidine on plasma catecholamine levels, vital signs such as systemic blood pressure, heart rate and sedation. The investigators will also monitor the local and systemic safety and tolerability of subcutaneously administered dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* Fluent skills in the Finnish language in order to be able to give informed consent and communicate with the study personnel.
* Age ≥ 18 years.
* Male gender.
* Weight ≥ 60 kg.
* Written informed consent from the subject.

Exclusion Criteria:

* Previous history of intolerance to the study drug or related compounds and additives.
* Concomitant drug therapy of any kind except paracetamol in the 14 days prior to the study.
* Existing or recent significant disease.
* History of any kind of drug allergy.
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements.
* Donation of blood within six weeks prior to and during the study.
* Body weight < 60 kg or BMI > 30 kg / m2.
* Participation in any other clinical study involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study.
* Smoking during one month before the start of the study or during the study period.
* Clinically significant abnormal findings in physical examination, ECG or laboratory screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability (%) of subcutaneously given dexmedetomidine | 10 hours
  Noncompartmental analysis after non-linear mixed effects modelling.

SECONDARY OUTCOMES:
Change in hemodynamic parameter (blood pressure) | 10 hours
  More than 30% change from the baseline in the blood pressure (measured in mmHg)
Number of participants with adverse events as a measure of safety and tolerability | 7 days
Change in hemodynamic parameter (heart rate) | 10 hours
  More than 30% change from the baseline in the blood pressure (measured in beats/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Teijo I Saari, MD, PhD, Principal Investigator — Dept. Anaesthesiology and Intensive Care, University Of Turku
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Ashraf MW, Uusalo P, Scheinin M, Saari TI. Population Modelling of Dexmedetomidine Pharmacokinetics and Haemodynamic Effects After Intravenous and Subcutaneous Administration. Clin Pharmacokinet. 2020 Nov;59(11):1467-1482. doi: 10.1007/s40262-020-00900-3. PMID 32462542
- [Derived] Uusalo P, Al-Ramahi D, Tilli I, Aantaa RA, Scheinin M, Saari TI. Subcutaneously administered dexmedetomidine is efficiently absorbed and is associated with attenuated cardiovascular effects in healthy volunteers. Eur J Clin Pharmacol. 2018 Aug;74(8):1047-1054. doi: 10.1007/s00228-018-2461-1. Epub 2018 Apr 17. PMID 29666901